CLINICAL TRIAL: NCT03791489
Title: Feasibility Study of Multi-Treatment Posterior Nasal Nerve (PNN) Modulation for Treatment of Chronic Rhinitis
Brief Title: Multi-Treatment PNN Modulation for Chronic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arrinex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-0005
Record Dates: First submitted 2018-12-31; First posted 2019-01-02 (Actual); Results first posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Chronic Rhinitis

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, feasibility study of multi-treatment locations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active Treatment (Experimental): Cryotherapy of the posterior nasal nerve using the ClariFix device
  Interventions: Device: ClariFix

INTERVENTIONS:
Device: ClariFix — The ClariFix™ device (K162608) is an FDA 510(k) cleared Class II cryosurgical tool indicated for the destruction of unwanted tissue during surgical procedures, including in adults with chronic rhinitis.

SUMMARY:
Feasibility of treatment at multiple sites with the ClariFix cryoablation device for treatment of chronic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Presence of moderate to severe rhinorrhea symptoms and mild to severe nasal congestion symptoms for >3 months.
* Documented allergy test within the last 10 years that defines whether or not subject has allergies to perennial and seasonal allergens, or is willing to have one performed prior to study exit.
* Able to provide informed consent and willing to complete study activities and visits per protocol.

Exclusion Criteria:

* Clinically significant anatomic obstructions that limit access to the posterior nose.
* Prior sinus or nasal surgery that significantly alters the anatomy of the posterior nose.
* Moderate to severe ocular symptoms as determined.
* History of epistaxis in the past 3 months.
* History of rhinitis medicamentosa.
* Prior head or neck irradiation.
* Active or chronic nasal or sinus infection.
* Pregnant.
* Allergy or intolerance to anesthetic agent.
* Cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, Raynaud's disease, and/or, open and/or infected wounds at or near the target tissue.
* Currently participating in another clinical research study.
* Any physical condition that, in the investigator's opinion, would prevent adequate study participation or pose increased risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Yen, MD, Principal Investigator — Specialty Physician Associates
Locations (3):
- United States (3):
  - San Francisco Otolaryngology Medical Group, San Francisco, California
  - Bethlehem ENT, Bethlehem, Pennsylvania
  - Tracy Byerly, MD, Fredericksburg, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: 30 Days
Arm/Group | Active Treatment
Started | 30
Completed | 30
Not Completed | 0
Period: 90 Days (Primary Endpoint)
Arm/Group | Active Treatment
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Active Treatment
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30
Number with allergic rhinitis [Count of Participants; unit: Participants] | 11
Number with nonallergic rhinitis [Count of Participants; unit: Participants] | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Procedure-related Serious Adverse Events (SAEs) and/or Serious Adverse Device Effects (SADE)
Description: The outcome measure is the number of participants experiencing 1 or more SAEs/SADEs.
Time Frame: Study duration (90-days)
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment
Number analyzed (Participants) | 30
Participants | 0

2. Secondary Outcome: Pain Scores
Description: Tolerability of treatment as provided by the participant by verbal report of pain/discomfort during treatment and post treatment using an 11-point scale indicating pain intensity from 0 (no pain) to 10 (worst pain).
Time Frame: Day of treatment during procedure and for up to 1 hour post procedure
Population: All enrolled participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 30
score on a scale
  During treatment | 1.0 (1.95)
  Post treatment | 4.1 (3.87)

3. Secondary Outcome: Change From Baseline in the Reflective Total Nasal Symptom Score (rTNSS)
Description: The rTNSS is a validated patient-reported outcome measure consisting of 4 symptoms: rhinorrhea, nasal congestion, nasal itching, and sneezing. Each item is scored on a scale of 0 (no symptoms) to 3 (severe symptoms). The total rTNSS is the sum of the 4 symptom scores and has a possible range of 0 to 12 points. The change from baseline is calculated as the follow-up value minus the baseline value. Negative values indicate improved symptoms.
Time Frame: 30 and 90 days after treatment
Population: All enrolled participants with the applicable follow-up visit.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 30
score on a scale
  30-day follow-up | -3.5 [-5.0 to -2.0]
  90-day follow-up | -4.0 [-6.0 to -1.0]
Statistical Analysis 1: Comparison: Active Treatment; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change From Baseline in the Overall Nasal Obstruction Symptom Evaluation (NOSE) Score
Description: The NOSE survey is a patient-reported outcome measure consisting of 5 nasal symptoms: nasal congestion or stuffiness, nasal blockage or obstruction, trouble breathing through the nose, trouble sleeping, and unable to get enough air through the nose during exercise or exertion. Each symptom is scored using a 5-point scale of 0 (not a problem) to 4 (severe problem). The 5 symptom scores are summed and the total is multiplied by 5 to give a total score that ranges from 0 to 100, with higher scores indicating worse symptoms. The change from baseline is calculated as the follow-up value minus the baseline value. Negative values indicate improved symptoms.
Time Frame: 30 and 90 days after treatment
Population: All enrolled participants with the applicable follow-up visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment
Number analyzed (Participants) | 30
score on a scale
  30-day follow-up | -19.0 (28.3)
  90-day follow-up | -31.4 (34.4)
Statistical Analysis 1: Comparison: Active Treatment; Test type: Superiority; p < 0.03, t-test, 2 sided — Threshold for statistical significance = p<0.05

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the study duration of 90 day after the ClariFix procedure.
Arm/Group | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 22/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=30)
Headache (Nervous system disorders) | 12 (12)
Postprocedure pain/discomfort (Injury, poisoning and procedural complications) | 10 (10)
Palate numbness (Injury, poisoning and procedural complications) | 8 (8)
Nasal discharge (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03791489/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03791489/SAP_001.pdf